CLINICAL TRIAL: NCT07290192
Title: Comparison of Impact of Step Down Verses Step Back Preparation Technique of Root Canals on Post Operative Pain in Patients Having Pulp Necrosis
Brief Title: This Study Compares Two Different Ways of Cleaning and Shaping Root Canals During Root-canal Treatment: the Step-down Technique and the Step-back Technique. Iu Want to Find Out Which Method Causes Less Pain After the Procedure. Patients Will be Randomly Placed Into One of the Two Groups, Treated Wit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Post Graduate Medical Institute (AFPGMI), Rawalpindi (Other)
Responsible Party: Principal Investigator, Kokab Naeem, Dentist, Armed Forces Post Graduate Medical Institute (AFPGMI), Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RCT-2025-pain-02
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pulp Necrosis
Keywords: Post operative pain; Pulp necrosis; Step back technique; Step down technique
MeSH Terms: conditions — Dental Pulp Necrosis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step back technique of root canal Vs step down technique of root canal (Experimental): Arm 1: Step-Down Technique
  Arm Type: Experimental Arm Title: Step-Down Root Canal Preparation
  Arm Description:
  Participants in this arm will receive root canal preparation using the step-down technique, where shaping begins in the coronal portion of the canal and progresses toward the apex. This method is designed to improve irrigation and reduce debris extrusion.
  ---
  Arm 2: Step-Back Technique
  Arm Type: Experimental Arm Title: Step-Back Root Canal Preparation
  Arm Description:
  Participants in this arm will receive root canal preparation using the step-back technique, where shaping starts at the apical portion and moves step-by-step backward toward the coronal area using progressively larger files. This conventional method serves as the comparison technique.
  Interventions: Procedure: Step down technique
- Arm 1 Arm Type: Experimental Arm Title: Step-Down Preparation Technique Detailed Description: Pa (Experimental): Participants in arm 1 will receive root canal preparation using the step-down technique, where shaping begins at the coronal portion of the canal and gradually progresses toward the apex. This method is intended to improve irrigation, reduce debris extrusion, and potentially lower postoperative pain.
  Participants arm 2 will receive root canal preparation using the step-back technique, where shaping starts at the apical portion and moves stepwise toward the coronal area using progressively larger files. This conventional method serves as the comparator to evaluate differences in postoperative pain and treatment outcomes.
  Interventions: Procedure: Step down technique

INTERVENTIONS:
Procedure: Step down technique — Step-Down Root Canal Preparation Experimental Step-Down Technique Procedure Root canal preparation starts at the coronal portion of the canal and progresses toward the apex using endodontic files of decreasing size. Aims to improve irrigation, reduce debris extrusion, and minimize postoperative pain.
  Step-Back Root Canal Preparation Active Comparator Step-Back Technique Procedure Root canal preparation starts at the apical portion of the canal and progresses stepwise toward the coronal portion using progressively larger files. Serves as the conventional comparator technique to evaluate postoperative pain

SUMMARY:
This randomized clinical trial aims to compare the step-back and step-down root canal preparation techniques in patients with pulp necrosis. The study will evaluate which technique results in less postoperative pain. Participants will be randomly assigned to one of the two groups. Pain intensity will be recorded at specific time points after the procedure using a standardized pain scale. The goal is to identify the technique that provides better patient comfort after root canal treatment.This study is a randomized clinical trial designed to compare the effects of two root canal preparation techniques-step-back and step-down-on postoperative pain in patients diagnosed with pulp necrosis. Participants will be randomly assigned to one of the two groups.

DETAILED DESCRIPTION:
This study is a randomized clinical trial designed to compare the effects of two root canal preparation techniques-step-back and step-down-on postoperative pain in patients diagnosed with pulp necrosis. Participants will be randomly assigned to one of the two groups.

In the step-down group, root canal shaping will begin at the coronal portion and gradually progress toward the apex, while in the step-back group, preparation will start at the apical portion and move backward toward the coronal area. Postoperative pain will be assessed at multiple time points using a standardized pain scale (e.g., Visual Analog Scale).

The aim of the study is to determine which technique causes less pain after treatment, helping clinicians choose the method that improves patient comfort following root canal therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients age between 18 to 65 years Healthy patients with ASA classification 1 and 2 Patients of both genders Patients who agreed to attend recall appointments Patients having single rooted tooth with pulp necrosis without pre-existing periapical pathosis and apical periodontitis

Exclusion Criteria:

* Patients with history of chronic pain Previously RCT treated tooth Teeth with apical pathosis ,with irreversible pulpitis Patients having systemic illness Multirooted teeth Patients consumed analgesics between appointments Teeth with calcified canals Cases of root fracture Children Pregnant and lactating mothers Smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain in patients undergoing root canal treatment using two techniques step back and step down in patients having pulp necrosis | 6 months of duration
  Patients randomly assigned in two groups Group A patients in which root canal treatment is done using step back technique Group B patients in which root canal treatment is done using step down technique Pain is assessed using visual analog scale ranging from 0(no pain) to 10 worst pain possible.Patients record their pain at 12,24,48 72 hours.Pain diaries will be collected at one week follow up.Data will be used to compare mean VAS between groups to evaluate the efficacy of two techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- Armed forces post graduate medical institute Rawalpindi ,Punjab Pakistan 46000, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participation data will not be shared because the study doesn't include plans or infrastructure for long term data storage de- identification and controlled access is needed to protect the participants privacy.Additionally the data set is small and disclosure may increase the risk of reidentification.Summary results will be made available as required .

REFERENCES:
- See also: Related Info — https://www.cureus.com/articles/169766-evaluation-of-the-impact-of-different-instrumentation-techniques-on-the-incidence-of-postoperative-pain-in-patients-undergoing-root-canal-treatment